CLINICAL TRIAL: NCT02321124
Title: Connective Tissue Manipulation Improves Symptoms and Quality of Life in Patients With Chronic Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceren Gürşen, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hacettepe University
Record Dates: First submitted 2014-12-09; First posted 2014-12-22 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Chronic Constipation
Keywords: Constipation; connective tissue manipulation; conservative therapy; massage; randomized controlled trial
MeSH Terms: conditions — Constipation

ARMS (2):
- intervention (Active Comparator): we will apply connective tissue manipulation and life style advice.
  Interventions: Other: connective tissue manipulation; Behavioral: life style advice
- control group (Other): We will apply only life style advice.
  Interventions: Behavioral: life style advice

INTERVENTIONS:
Other: connective tissue manipulation — We will apply connective tissue manipulation 5 days a week for four weeks.
  Arms: intervention
Behavioral: life style advice — We will apply life style advice for four weeks.

SUMMARY:
Connective tissue manipulation (CTM) is a manual reflex therapy, which increases intestinal motility by stimulating autonomic nervous system to re-balance the parasympathetic and sympathetic functions. However, there is no randomized controlled trial (RCT) regarding the efficacy of CTM on constipation. This study was planned to investigate the effects of CTM in patients with chronic constipation.

Patients who have diagnosis of chronic constipation according to Rome III criteria were recruited and randomized to intervention and control group. The intervention group received CTM in addition to the lifestyle advice, while the control group was given only lifestyle advice for constipation. All assessments were performed at baseline and at the end of 4 weeks. The primary outcome measure was the Constipation Severity Instrument (CSI). Secondary outcomes included Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL), Bristol Stool Scale (BSS) and 7-day bowel diary. Differences between groups were analyzed with t-tests, Mann-Whitney U test and Chi-square test.

DETAILED DESCRIPTION:
In this prospective randomized controlled trial, informed consent forms were obtained from all participants and they were informed about the study based on the Declaration of Helsinki. The study was approved by local ethics committee of Hacettepe University (LUT 12/35-48). After comprehensive clinical evaluation, subjects were randomly assigned to the intervention group or the control group, using stratified block randomization procedure with blocks of four, using opeque and sealed envelopes, containing group allocation number from a computer generated random number table The intervention group received CTM in addition to the lifestyle advice, while the control group was given only lifestyle advice for constipation.

Patients diagnosed with chronic constipation by a based on Rome III Criteria were recruited by a gastroenterologist from Hacettepe University, Adult Hospital, Gastroenterology Unit and the patients were evaluated and treated at Hacettepe University, Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Women's Health Unit.

Participants were recruited if they were over 18 years of age and had a diagnosis of chronic constipation according to Rome III criteria. Exclusion criteria were comorbid neurological, anatomical, or metabolic condition, pregnancy, mental problems preventing cooperation, history of colostomy surgery, history of gastrointestinal, spinal, or pelvic surgery except cholecystectomy, appendectomy, or hysterectomy, comorbid various colonic conditions (intestinal obstruction, peritonitis, bowel perforation, peptic ulcer, gastrointestinal bleeding, or acute inflammation of abdominal organs), history of intestinal cancer, existence of open sore or tumor at the massage region, and abdominal hernia. Patients taking laxatives were excluded or were asked to discontinue the drug two weeks before enrollment.

Intervention CTM was applied five days per week, a total of 20 sessions for 4 weeks. Each session lasted around 15-20 minutes. While patients were in a sitting position, starting from the lumbosacral region, lower thoracic, scapular, inter-scapular and cervical regions were included in the treatment, respectively. All patients were also advised to increase their physical activity levels, fluid and fibre intake, and to take the ideal posture for defecation (squatting position) with a two-pages document.

Evaluations Physical (age, gender, Body Mass Index (BMI)(kg/m²) and demographic (educational status, duration of constipation, marital status, employment status) data of the participants were recorded. In addition, the number of meals per day, daily amount of liquid consumption, and physical activity levels were recorded. The participants' physical activity levels were measured using the Turkish version of the International Physical Activity Questionnaire-Short Form (IPAQ-SF). Measurements were performed at baseline and immediately after the treatment. All patients were evaluated by the same experienced therapist, who was blinded to the results of the pre-treatment measurements (CG).

The primary outcome measure

*Constipation Severity Instrument (CSI) To evaluate the severity of the participants' constipation, Constipation Severity Instrument (CSI) was used. CSI was designed to evaluate individuals' defecation frequency and consistency as well as the level of straining experienced by individuals during bowel movement. There are three subscales of CSI, obstructive defecation (OT), colonic inertia (CI), and pain. Higher scores of CSI indicate more severe constipation. Kaya et al. showed that the Turkish version of CSI is reliable and valid in determining constipation and grading of its severity.

Secondary outcome measures

* Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL) Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL) includes a total of 28 items in 4 subscales: worries and concerns (11 items), physical discomfort (4 items), psychosocial discomfort (8 items), and satisfaction (5 items). Higher scores of PAC-QOL indicate more negative effects of constipation on the quality of life. Turkish version of PAC-QOL was demonstrated to be reliable and valid.
* Bristol Stool Scale (BSS) The stool consistency was evaluated using the Bristol Stool Scale (BSS), a seven-point scale (from 1 to 7), where 1 =separate hard lumps, like nuts; 2=sausage shaped but lumpy; 3 = like a sausage or snake, but with cracks on its surface; 4 = like a sausage or snake, smooth and soft; 5 = soft blobs with clear cut edges; 6=ﬂuffy pieces with ragged edges, a mushy stool; 7=water, no solid pieces.
* 7-Day Bowel Diary In order to gather information regarding the participants' symptoms of constipation, they were asked to complete a 7-day bowel diary before and after the treatment. This diary included items regarding the frequency of bowel movement, stool consistency, defecation time, feeling of incomplete evacuation, and changes in food and liquid consumption.
* Perception of Subjective Change Individuals' perception of subjective change after the treatment was evaluated using a 5-point Likert-type scale: 0: No change, 1: Minimal change, 2: Moderate change, 3: Important change, 4: Very important change.
* Compliance to the Advices Compliance of the participants to lifestyle advices was evaluated using a 4-point Likert-type scale: 0: No compliance, 1: minimal compliance, 2: moderate compliance, and 3: Full compliance.

ELIGIBILITY:
Inclusion Criteria:

* Participants were recruited if they were over 18 years of age and had a diagnosis of chronic constipation according to Rome III criteria.

Exclusion Criteria:

* Exclusion criteria were comorbid neurological, anatomical, or metabolic condition, pregnancy, mental problems preventing cooperation, history of colostomy surgery, history of gastrointestinal, spinal, or pelvic surgery except cholecystectomy, appendectomy, or hysterectomy, comorbid various colonic conditions (intestinal obstruction, peritonitis, bowel perforation, peptic ulcer, gastrointestinal bleeding, or acute inflammation of abdominal organs), history of intestinal cancer, existence of open sore or tumor at the massage region, and abdominal hernia. Patients taking laxatives were excluded or were asked to discontinue the drug two weeks before enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Constipation Severity Instrument (CSI) | Participants will be followed for four weeks. Change from baseline severity of constipation at 4 weeks will be evaluated.
  Constipation Severity Instrument was designed to evaluate individuals' defecation frequency and consistency as well as the level of straining experienced by individuals during bowel movement. There are three subscales of CSI, obstructive defecation (OT), colonic inertia (CI), and pain. Higher scores of CSI indicate more severe constipation.

SECONDARY OUTCOMES:
Patient-Assessment of Quality of Life Questionnaire (PAC-QOL) | Participants will be followed for four weeks. Change from baseline quality of life at 4 weeks will be assessed.
  Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL) includes a total of 28 items in 4 subscales: worries and concerns (11 items), physical discomfort (4 items), psychosocial discomfort (8 items), and satisfaction (5 items).
Bristol Stool Scale | Participants will be followed for four weeks. Change from baseline stool consistency at 4 weeks will be assessed.
  The stool consistency was evaluated using the Bristol Stool Scale (BSS), a seven-point scale (from 1 to 7), where 1 =separate hard lumps, like nuts; 2=sausage shaped but lumpy; 3 = like a sausage or snake, but with cracks on its surface; 4 = like a sausage or snake, smooth and soft; 5 = soft blobs with clear cut edges; 6=ﬂuffy pieces with ragged edges, a mushy stool; 7=water, no solid pieces.
7-day bowel diary | Participants will be followed for four weeks. Change from baseline symptoms of constipation at 4 weeks will be evaluated.
  This diary included items regarding the frequency of bowel movement, stool consistency, defecation time, feeling of incomplete evacuation, and changes in food and liquid consumption.
perception of subjective change | Participants will be followed for four weeks. Change of subjective change from baseline after 4 week treatment will be assessed.
  Individuals' perception of subjective change after the treatment was evaluated using a 5-point Likert-type scale: 0: No change, 1: Minimal change, 2: Moderate change, 3: Important change, 4: Very important change.
compliance with advice | Participants will be followed for four weeks. Change of compliance with advice from baseline after 4 week treatment will be assessed.
  Compliance of the participants to lifestyle advices was evaluated using a 4-point Likert-type scale: 0: No compliance, 1: minimal compliance, 2: moderate compliance, and 3: Full compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Gursen, Principal Investigator — Hacettepe University; Mintaze Kerem Gunel, Study Director — Hacettepe University; Serap Kaya, Principal Investigator — Hacettepe University; Taylan Kav, Study Director — Hacettepe University; Türkan Akbayrak, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Holey EA, Lawler HL. The effects of classical massage and connective tissue manipulation on bowel function. Br J Ther Rehabil 1995;211:627-31.
- [Background] Quist DM, Duray SM. Resolution of symptoms of chronic constipation in an 8-year-old male after chiropractic treatment. J Manipulative Physiol Ther. 2007 Jan;30(1):65-8. doi: 10.1016/j.jmpt.2006.11.005. PMID 17224358
- [Background] Simmons SF, Schnelle JF. Effects of an exercise and scheduled-toileting intervention on appetite and constipation in nursing home residents. J Nutr Health Aging. 2004;8(2):116-21. PMID 14978607
- [Background] Holey LA, Dixon J. Connective tissue manipulation: a review of theory and clinical evidence. J Bodyw Mov Ther. 2014 Jan;18(1):112-8. doi: 10.1016/j.jbmt.2013.08.003. Epub 2013 Sep 8. PMID 24411158
- See also: rome foundation — http://www.romecriteria.org